CLINICAL TRIAL: NCT04672863
Title: Effects of a Structured, Modified Mediterranean Dietary Intervention After Liver Transplantation
Brief Title: Mediterranean Diet Post-liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kymberly D. Watt, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-009762
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (No Intervention): Subjects will participate in a standardized Transplant Nutrition class between day 21-40 as per institutional protocol and will be counseled as per the Mayo Clinic standard of care vis a vis dietary intervention, standard aerobic and resistance exercise recommendations (consistent with AASLD guidelines) and other lifestyle interventions.
- Behavioral: Structured Modified Mediterranean Diet (Experimental): Subjects will participate in a one-on-one counselling session with a dietician, as opposed to attending the standardized Transplant Nutrition class. Counselling will be provided on the elements of the modified Mediterranean diet which emphasizes consumption of fruits, vegetables, whole grains, beans and nuts, in addition to low salt, moderate amounts of lean protein (primarily fish and poultry) in addition to low to moderate quantities of monounsaturated fats.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — Modified Mediterranean diet approved by the Nutrition Team at the Transplant Center and it emphasizes consumption of fruits, vegetables, whole grains, beans and nuts, in addition to low salt (2-2.4g/day), moderate amounts of lean protein (primarily fish and poultry) in addition to low to moderate quantities of monounsaturated fats. The modifications to the traditional Mediterranean diet are: no alcohol consumption and fewer added fats. In addition, close scheduled followup on diet and progress with study team.
  Arms: Behavioral: Structured Modified Mediterranean Diet

SUMMARY:
The purpose of this study is to study the effects of a structured Mediterranean dietary program on prevention of weight gain, promotion of heart health and prevention of fatty liver disease after liver transplantation.

DETAILED DESCRIPTION:
Study Hypotheses

* A modified Mediterranean diet after liver transplantation results in weight loss, improvement of insulin sensitivity, lipid profiles, blood pressure, BMI, and waist circumference in patients who adhere to the program.
* A modified Mediterranean diet after liver transplantation results in relative improvement in cardiovascular outcomes in patients who adhere to the program when compared to standard of care.
* A modified Mediterranean diet after liver transplantation results in relative improvement in 10-year ASCVD risk in patients who adhere to the program when compared to standard of care.
* A modified Mediterranean diet after liver transplantation decreases the risk of development of NAFLD/NASH/NASH fibrosis in patients who adhere to the program.

Study Design:

* Single-center, prospective, randomized interventional trial
* All eligible post-liver transplant patients during the enrollment period will be invited to participate in the trial.
* All enrolled patients will be randomized to the Dietary Intervention (DI) arm or the Standard of Care (SOC) arm.
* All patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria

* Adult patients ≥ 18 years of age undergoing primary liver transplant
* Ascites-adjusted BMI ≥ 25 kg/m2
* Acceptable graft function (total bilirubin level < 5 mg/dL and doppler ultrasound with patent hepatic artery, hepatic veins and portal veins)

Exclusion Criteria

* Hepatocellular carcinoma (HCC) that did not fulfill Milan criteria as per explant histology
* Untreated post-transplant vascular complications or biliary strictures
* Multi-organ transplantation
* Urine protein excretion ≥2.0 g/day
* Uncontrolled diabetes mellitus (HbA1c > 10%)
* Associated medical conditions incompatible with safe participation in a nutritional intervention study, including digestive diseases with fat intolerance, neurological, psychiatric or endocrine disorders
* Active eating disorder (e.g. bulimia nervosa, anorexia nervosa)
* History of bariatric surgery
* Pregnancy or planning on pregnancy in the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
weight gain | 4 months
  weight in kilograms
weight gain | 12 months
  weight in kilograms

SECONDARY OUTCOMES:
fat mass changes | 4 months
  InBody body composition analysis of fat mass vs lean body mass changes
fat mass changes | 12 months
  InBody body composition analysis of fat mass vs lean body mass changes

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly Watt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials